CLINICAL TRIAL: NCT06900166
Title: A Prospective, Open-Label, Randomized, Controlled, Multicenter Clinical Study of Pegylated Interferon Alfa-2b in Reducing Relapse Rates After Nucleos(t)ide Analogue Withdrawal in HBeAg-Negative Chronic Hepatitis B Patients with Low-Level HBsAg
Brief Title: Pegylated Interferon Alfa-2b in Reducing Relapse Rates After Nucleos(t)ide Analogue Withdrawal in HBeAg-negative CHB Patients with Low Level HBsAg
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jiming Zhang, chief physician,professor, Huashan Hospital
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEASE2.0
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Nucleobindins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Controlled Group (No Intervention): Directly stopped NUC, follow-up to 96 weeks
- PegIFN alfa-2b 48 weeks (Active Comparator): Discontinue the NUC treatment ,PegIFN alfa-2b for 48 weeks and follow up for 96 weeks
  Interventions: Drug: PegIFN alfa-2b
- PegIFN alfa-2b and NUC 48 weeks (Experimental): Discontinue the NUC treatment ,PegIFN alfa-2b and NUC for 48 weeks, then follow up for 96 weeks
  Interventions: Drug: PegIFN alfa-2b and NUC

INTERVENTIONS:
Drug: PegIFN alfa-2b — 180 μg/ 0.5 ml ,hypodermic injection once a week
  Arms: PegIFN alfa-2b 48 weeks
Drug: PegIFN alfa-2b and NUC — 180 μg/ 0.5 ml ,hypodermic injection once a week, NUC drugs should be used according to the instructions of each drug
  Arms: PegIFN alfa-2b and NUC 48 weeks

SUMMARY:
All enrolled patients must meet the European Guidelines for the Prevention and Treatment of Chronic Hepatitis B (EASL, 2017) recommended discontinuation criteria, that is, HBeAg-negative chronic hepatitis B patients without fibrosis or cirrhosis who have undetectable HBV DNA for more than 3 years after receiving NUC treatment can attempt to discontinue the drug. At the same time, the patient's HBsAg level will not be higher than 1000 IU/mL. The study will set up three groups, group A directly stopped nucleoside analogues, follow-up to 96 weeks; Group B received PegIFNα-2b monotherapy for 48 weeks, group C received PegIFNα-2b combined with NUC treatment for 48 weeks, group B and group C stopped all antiviral drugs after completing 48 weeks of treatment, and then followed up for 96 weeks, a total of 144 weeks of follow-up. This study aims to further optimize the design on the basis of previous clinical studies to observe whether sequential interferon or combined with NUC therapy can reduce the virological relapse rate of HBeAg-negative chronic hepatitis B patients with low HBsAg level after 96 weeks of discontinuation, and to observe the impact on the functional cure rate.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 65 (inclusive), regardless of gender;
2. Fibroscan ≤ 7.4kpa;
3. HBeAg-negative CHB patients: HBsAg positive, HBeAg negative, HBsAb negative and HBeAb positive before receiving NUC treatment and during screening in this study;
4. HBeAg-negative chronic hepatitis B patients without liver cirrhosis who have been viral-negative for more than 3 years after receiving NUC treatment, and they meet the 2017 EASL guideline discontinuation standard (HBV DNA is lower than the lower limit of detection, that is, <20 IU/ml);
5. HBsAg≤1000 IU/ml;
6. Have the intention to stop taking the drug, and sign a written informed consent.

Exclusion Criteria:

1. HBsAb positive during screening;
2. Patients with hepatitis B cirrhosis in the compensatory and decompensated stage: patients with a clear history of cirrhosis (imaging or histological evidence) or Child-Pugh score ≥5 before NUC treatment, or complications of cirrhosis in the decompensated stage such as ascites, hepatic encephalopathy, esophageal variceal hemorrhage, etc.;
3. Patients who are allergic to alpha interferon and its drug ingredients, and the researchers judge that alpha interferon is not suitable for patients;
4. Received immunomodulators (including interferon, etc.) within 1 year before screening;
5. Combined with HAV, HCV, HDV, HEV, HIV infection, alcoholic liver disease, genetic metabolic liver disease, drug liver disease, non-alcoholic fatty liver disease and other chronic liver diseases;
6. Combined with autoimmune diseases, including autoimmune liver disease, psoriasis, etc.
7. Patients with primary liver cancer or screening with AFP greater than 100 ng/ml and imaging findings indicating the possibility of malignant liver occupation; Or AFP greater than 100 ng/ml for 3 months;
8. Neutrophil count < 1.5 x 109 cells /L or platelet count < 90 x 109 cells /L;
9. Creatinine is 1.5 times higher than the upper limit of normal;
10. Patients with other malignant tumors (excluding cured patients);
11. Patients with serious diseases of heart, lung, kidney, brain, blood and other important organs;
12. Patients with severe neurological and psychiatric disorders (such as epilepsy, depression, mania, seizures, schizophrenia, etc.);
13. Control unstable diabetes, hypertension, thyroid disease, etc.;
14. Pregnant and lactating women or patients who had pregnancy plans during the study period and did not want to use contraception;
15. Participate in other clinical investigators;
16. Patients who were not considered suitable for participation in this study by the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants who relapse | 96 weeks after stopping NAs
  the cumulative virological relapse rate (HBV DNA>2000 IU/ml on 2 separate occasions 1 months apart) during the research period.

SECONDARY OUTCOMES:
Number of participants who relapse | 72 weeks after stopping all antivirals
  The total number of relapse (HBV DNA>2000 IU/ml on 2 separate occasions 1 months apart) during the research period.
Number of participants who relapse Clinically | 72 weeks and 96 weeks after stopping all antivirals
Number of participants who achieve HBsAg clearance and HBsAg seroconversion | 96 weeks after stopping all antivirals
Number of participants who restart treatment | 96 weeks after stopping all antivirals
  Patients with virological relapse may be retreated according to the following criteria: 1) ALT >10×ULN, 2)ALT >5×ULN and total bilirubin >2 mg/dl, 3)ALT >3×ULN and HBV DNA >100,000 IU/ml, 4) ALT >ULN and HBV DNA >2,000 IU/ml for more than 3 months; 5) PT increases by more than 2s, while ALT >5×ULN.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator Jiming Zhang, M.D., Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Papatheodoridi M, Papachristou E, Moschidis Z, Hadziyannis E, Rigopoulou E, Zachou K, Villeret F, Magiorkinis G, Lyberopoulou A, Gatselis N, Vlachogiannakos I, Manolakopoulos S, Dalekos GN, Zoulim F, Paraskevis D, Papatheodoridis GV. Significance of serum HBV RNA in non-cirrhotic HBeAg-negative chronic hepatitis B patients who discontinue effective antiviral therapy. J Viral Hepat. 2022 Nov;29(11):948-957. doi: 10.1111/jvh.13729. Epub 2022 Aug 30. PMID 35789515
- [Background] Hirode G, Choi HSJ, Chen CH, Su TH, Seto WK, Van Hees S, Papatheodoridi M, Lens S, Wong G, Brakenhoff SM, Chien RN, Feld J, Sonneveld MJ, Chan HLY, Forns X, Papatheodoridis GV, Vanwolleghem T, Yuen MF, Hsu YC, Kao JH, Cornberg M, Hansen BE, Jeng WJ, Janssen HLA; RETRACT-B Study Group. Off-Therapy Response After Nucleos(t)ide Analogue Withdrawal in Patients With Chronic Hepatitis B: An International, Multicenter, Multiethnic Cohort (RETRACT-B Study). Gastroenterology. 2022 Mar;162(3):757-771.e4. doi: 10.1053/j.gastro.2021.11.002. Epub 2021 Nov 9. PMID 34762906
- [Background] Hall SAL, Burns GS, Anagnostou D, Vogrin S, Sundararajan V, Ratnam D, Levy MT, Lubel JS, Nicoll AJ, Strasser SI, Sievert W, Desmond PV, Ngu MC, Angus P, Sinclair M, Meredith C, Matthews G, Revill PA, Jackson K, Littlejohn M, Bowden DS, Locarnini SA, Visvanathan K, Thompson AJ. Stopping nucleot(s)ide analogues in non-cirrhotic HBeAg-negative chronic hepatitis B patients: HBsAg loss at 96 weeks is associated with low baseline HBsAg levels. Aliment Pharmacol Ther. 2022 Jul;56(2):310-320. doi: 10.1111/apt.16968. Epub 2022 May 6. PMID 35521992
- [Background] Liaw YF, Kao JH, Piratvisuth T, Chan HL, Chien RN, Liu CJ, Gane E, Locarnini S, Lim SG, Han KH, Amarapurkar D, Cooksley G, Jafri W, Mohamed R, Hou JL, Chuang WL, Lesmana LA, Sollano JD, Suh DJ, Omata M. Asian-Pacific consensus statement on the management of chronic hepatitis B: a 2012 update. Hepatol Int. 2012 Jun;6(3):531-61. doi: 10.1007/s12072-012-9365-4. Epub 2012 May 17. PMID 26201469
- [Background] European Association For The Study Of The Liver. EASL clinical practice guidelines: Management of chronic hepatitis B virus infection. J Hepatol. 2012 Jul;57(1):167-85. doi: 10.1016/j.jhep.2012.02.010. Epub 2012 Mar 20. No abstract available. PMID 22436845
- [Background] Lok AS, McMahon BJ. Chronic hepatitis B: update 2009. Hepatology. 2009 Sep;50(3):661-2. doi: 10.1002/hep.23190. No abstract available. PMID 19714720